CLINICAL TRIAL: NCT02541877
Title: A Prospective, Multi-center,Randomized Controled Trial of Sizing-strategy of Bicuspid Aortic Valve Stenosis With Transcatheter Self-expandable Valve
Brief Title: Sizing-sTrategy of Bicuspid AoRtic Valve Stenosis With Transcatheter Self-expandable Valve
Acronym: START
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jian'an Wang,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZJU CT004
Record Dates: First submitted 2015-08-14; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Down sizing valve in type-0 BAS (Experimental): Down Sizing Transcatheter Self-expandable Valve in Type-0 BAS
  Interventions: Device: Down sizing valve in type-0 BAS
- Standard sizing valve in type-0 BAS (Active Comparator): Standard Sizing Transcatheter Self-expandable Valve in Type-0 BAS
  Interventions: Device: Standard sizing valve in type-0 BAS
- Standard sizing valve in TAS (Active Comparator): Standard Sizing Transcatheter Self-expandable Valve in TAS
  Interventions: Device: Standard sizing valve in TAS

INTERVENTIONS:
Device: Down sizing valve in type-0 BAS — Subjects will undergo percutaneous retrograde trans-peripheral arterial aortic valve implantation with the self-expandable bio-prosthesis. Before implantation a balloon dilatation of the aortic annulus and a simultaneous aortic root angiography will be performed. Down sizing valve implantation will be used in type-0 BAS.
  Arms: Down sizing valve in type-0 BAS
Device: Standard sizing valve in type-0 BAS — Subjects will undergo percutaneous retrograde trans-peripheral arterial aortic valve implantation with the self-expandable bio-prosthesis. Before implantation a balloon dilatation of the aortic annulus and a simultaneous aortic root angiography will be performed. Standard sizing valve implantation will be used in type-0 BAS.
  Arms: Standard sizing valve in type-0 BAS
Device: Standard sizing valve in TAS — Subjects will undergo percutaneous retrograde trans-peripheral arterial aortic valve implantation with the self-expandable bio-prosthesis. Before implantation a balloon dilatation of the aortic annulus and a simultaneous aortic root angiography will be performed. Standard sizing valve implantation will be used in TAS.
  Arms: Standard sizing valve in TAS

SUMMARY:
To observe the clinical outcomes of the different valve sizing strategies treating type-0 Bicuspid Aortic Stenosis (BAS) with self-expandable transcatheter aortic valve implantation (TAVI) valve, compared with those of a standard sizing strategy of normal Tricuspid Aortic Stenosis(TAS).

DETAILED DESCRIPTION:
BACKGROUND: From our current clinical experience, investigators mostly choose the smaller self-expandable transcatheter valve for type-0 BAS than that for TAS, combined with "balloon sizing" strategy. But no prospective and randomized studies show the rationality and clinical outcomes of different sizing strategies of type-0 BAS with self-expandable transcatheter valve.

AIM: To observe the clinical outcomes of the different valve sizing strategies treating type-0 BAS with self-expandable transcatheter aortic valve implantation (TAVI) valve, compared with those of a standard sizing strategy of normal TAS.

POPULATION: All patients with severe degenerative aortic valve stenosis referred for aortic valve intervention will be screened for study eligibility. To be included subjects must be 65 years or older, anatomical and technical eligible for both interventions, expected to survive more than 1 year after the intervention, and able to provide written informed consent. Study exclusion criteria include isolated aortic valve regurgitation or other significant valve disease, unstable preoperative condition.

DESIGN: The project is a multicenter randomized clinical trial. Patients of type-0 BAS fulfilling all inclusion and no exclusion criteria will be randomized into either Down sizing group or Standard sizing group. Randomization will be 1:1 with 53 subjects in each group. Meanwhile patients of TAS fulfilling all inclusion and no exclusion criteria will be included as a Standard group in this study. Screening and inclusion will commence in September 2015. Inclusion is expected to last 3 years, and subjects will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic severe aortic stenosis (echocardiographic criteria: AV effective orifice area (EOA) of < 1 cm2, mean AV gradient of > 40 mmHg, or AV peak systolic velocity of > 4.0 m/s; NYHA-class II or greater, angina pectoris, or syncope)
2. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
3. The subject agrees to comply with specified follow-up evaluations and to return to the investigational site where the procedure was performed.
4. Patients are technical and anatomical eligible for interventions

Exclusion Criteria:

1. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

   * Aspirin
   * Heparin (HIT/HITTS) and bivalirudin
   * Nitinol (titanium or nickel)
   * Ticlopidine and clopidogrel
   * Contrast media
2. Subject refuses a blood transfusion.
3. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
4. Native aortic annulus size < 20 mm or > 29 mm per the baseline diagnostic imaging.
5. Life expectancy is less than one year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Device success | At 24 hours after procedure
  1. Absence of procedural mortality
  2. Correct positioning of a single prosthetic heart valve into the proper anatomical location
  3. Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation)
Changes of prosthetic valve functions | From 24 hours after procedure to 5 years
  1. Valve hemodynamics
  2. Peri-valvular regurgitation
  3. Valve malpositioning
  4. Valve morphology

SECONDARY OUTCOMES:
All-cause mortality and all stroke (disabling and non-disabling) | 5 years
Number of patients with procedural complications | Within first 30 days
Changes of ascending aortic diameter | Changes of baseline ascending aortic diameter at 5 years
Functional status (NYHA-classification) | 5 years
Quality of Life (SF-12) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China